CLINICAL TRIAL: NCT02842762
Title: The Hemodynamic Effect of Transient Epicardial Right Ventricular Pacing After Cardiopulmonary Bypass, Assessed by Real-time Three-dimensional Echocardiography.
Brief Title: 3D Echocardiographic Assessment of Epicardial Pacing After Cardiopulmonary Bypass.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suzanne Flier, MD (Other)
Responsible Party: Sponsor-Investigator, Suzanne Flier, MD, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 108176
Record Dates: First submitted 2016-07-20; First posted 2016-07-25 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Disorder of Pacing Function
Keywords: Echocardiography, Three-dimensional; Cardiac Surgical Procedures; Cardiac Pacing, Artificial; Anesthesia
MeSH Terms: interventions — Cardiac Surgical Procedures; Device Lead Extraction

STUDY DESIGN:
Intervention Model Description: Sequence of measurements, during sinus rhythm and during pacing is randomized.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-paced (Sham Comparator): * cardiac surgery
  * 3D TEE measurements of systolic dyssynchrony
  * right ventricular epicardial pacemaker lead (off)
  Interventions: Procedure: cardiac surgery; Device: 3D TEE; Device: Pacemaker lead
- Paced (Experimental): The patient is randomized to the order of measurements taken, and serves as his own control.
  * cardiac surgery
  * 3D TEE measurements of systolic dyssynchrony
  * right ventricular epicardial pacemaker lead (on)
  Interventions: Device: Right ventricular epicardial pacing; Procedure: cardiac surgery; Device: 3D TEE; Device: Pacemaker lead

INTERVENTIONS:
Device: Right ventricular epicardial pacing — The patient's own heart rate at that moment will be the starting point for the study. Right ventricle pacing will be instituted by selecting a rate that is 5 beats above the patient's own heart rate. We will use a stepwise approach where we increase the pacermaker's rate with steps of 5 beats until we have 100% capture of the pacemaker beats. After waiting for at least one minute of pacing we will obtain a set of measurements.
  Arms: Paced
Procedure: cardiac surgery — Elective cardiac surgery, with use of cardiopulmonary bypass.
Device: 3D TEE — Intraoperatively, all patients will be monitored by means of TEE
  Other Names: three-dimensional transesophageal echocardiography
Device: Pacemaker lead — All patients will have a epicardial pacemaker lead in situ.

SUMMARY:
This study evaluates the usefulness of 3D echocardiography to guide pacemaker therapy in the operating room in cardiac surgical patients. Each patient will serve as his own control, following a paired design.

DETAILED DESCRIPTION:
Cardiac surgical patients sometimes require temporary pacing wires to optimize cardiac function during weaning from cardiopulmonary bypass (CPB), and/or to treat hemodynamically significant brady-arrhythmias. The available patient series report that 8.6% to 23.9% of patient undergoing coronary artery bypass grafting (CABG) or valve surgery require temporary pacing at some time after CPB. The site of pacemaker wire placement seems to be a crucial determinant of cardiac output. In non-surgical patients isolated right ventricular (RV) pacing seems to induce electromechanical dyssynchrony of the RV and the left ventricle (LV). A normal ventricle in sinus rhythm displays a simultaneous contraction of all segments of the heart, so that regional minimal volume (i.e. maximal contraction) will occur at the same time. Isolated RV pacing seems to result in a left bundle branch type electrical activation sequence, with delayed contraction of some of the segments. The LV, but not the RV, seems to negatively affected by this state of dyssynchrony, resulting in decreased cardiac output. In surgical patients however, there is not such data available yet. Since isolated RV epicardial wire placement is still widely practiced in cardiac surgery, and in our own institution, we would like to study the effect of RV pacing on LV synchrony and LV output.

Again from studies in non-surgical patients receiving resynchronization therapy, we know that real-time three-dimensional (3D) echocardiography is very useful to pick up subtle changes in LV synchrony and thereby guide synchronization of ventricular contraction. However, to date the usefulness of real-time 3D echocardiography to guide pacemaker therapy in cardiac surgery is unknown. In the present feasibility study in cardiac surgical patients, we want to investigate the acute effects of isolated RV pacing on LV synchrony, and LV output.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient scheduled to undergo elective cardiac surgery by means of full sternotomy and use of cardiopulmonary bypass
* Preoperative moderate to good LV function, ejection fraction > 30%
* Age > 18 yrs. old
* Preoperative sinus rhythm
* Pacemaker lead inserted by cardiac surgeon during surgery
* Underlying sinus rhythm after cardiopulmonary bypass before the end of surgery
* Able to understand written and verbal patient information
* Signed informed consent

Exclusion Criteria:

* Emergency cardiac surgery
* Minimally invasive surgery
* Contraindication to TEE
* Redo surgery
* Hemodynamic instability after CPB (late exclusion criterium)
* No pacemaker lead inserted by cardiac surgeon (late exclusion criterium)
* No sinus rhythm during chest closure towards the end of surgery (late exclusion criterium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Left ventricular systolic dyssynchrony index (SDI) | Intraoperative, end of cardiac surgery (duration 10 minutes)
  For each segment of 16 segments excluding the apical cap in a standard 17-segment model, the time to reach regional minimal volume is calculated as a fraction of the total cardiac cycle (RR interval) and expressed as a percentage.10 The standard deviation of these measurements is defined as the SDI. Three-dimensional SDI is therefore the dispersion time to reach the minimum systolic volume (as recommended).

SECONDARY OUTCOMES:
Ventricular volumes and ejection fraction | Intraoperative, end of cardiac surgery (duration 10 minutes)
  We will obtain a full volume 3D dataset and obtain end diastolic (EDV) and end systolic volume (ESV). By subtracting ESV from EDV we will obtain the ejection fraction (EF).
LVOT blood flow | Intraoperative, end of cardiac surgery (duration 10 minutes)
  As a surrogate for cardiac output we will obtain the velocity time integral (VTI) across the left ventricular outflow tract (LVOT)
Presence and severity of mitral regurgitation | Intraoperative, end of cardiac surgery (duration 10 minutes)
  From midesophageal position we will perform a transesophageal echocardiography (TEE) study to interrogate the mitral valve for the presence and severity of mitral regurgitation.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Flier, MD MSc, Principal Investigator — London Health Sciences Center
Locations (1):
- University Hospital - London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolber T, Haegeli L, Huerlimann D, Brunckhorst C, Luscher TF, Duru F. Altered left ventricular contraction pattern during right ventricular pacing: assessment using real-time three-dimensional echocardiography. Pacing Clin Electrophysiol. 2011 Jan;34(1):76-81. doi: 10.1111/j.1540-8159.2010.02908.x. Epub 2010 Oct 14. PMID 20946287
- [Background] Kapetanakis S, Kearney MT, Siva A, Gall N, Cooklin M, Monaghan MJ. Real-time three-dimensional echocardiography: a novel technique to quantify global left ventricular mechanical dyssynchrony. Circulation. 2005 Aug 16;112(7):992-1000. doi: 10.1161/CIRCULATIONAHA.104.474445. Epub 2005 Aug 8. PMID 16087800
- [Background] Alwaqfi NR, Ibrahim KS, Khader YS, Baker AA. Predictors of temporary epicardial pacing wires use after valve surgery. J Cardiothorac Surg. 2014 Feb 12;9:33. doi: 10.1186/1749-8090-9-33. PMID 24521215
- [Background] Bethea BT, Salazar JD, Grega MA, Doty JR, Fitton TP, Alejo DE, Borowicz LM Jr, Gott VL, Sussman MS, Baumgartner WA. Determining the utility of temporary pacing wires after coronary artery bypass surgery. Ann Thorac Surg. 2005 Jan;79(1):104-7. doi: 10.1016/j.athoracsur.2004.06.087. PMID 15620924